CLINICAL TRIAL: NCT06645782
Title: Virtual, Group Adaptation of a Cystic Fibrosis (CF) Specific Cognitive Behavioural Therapy for Adults With CF: An Exploration of Effectiveness, Feasibility, and Participant Experiences.
Brief Title: Group Cognitive Behavioural Therapy for Adults With Cystic Fibrosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Principal Investigator, Anna Dollimount, Principal Investigator, University of Regina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-644
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis (CF)
Keywords: Cystic Fibrosis; Cognitive Behavioural Therapy; Group Therapy; Mental Health; Internet
MeSH Terms: conditions — Cystic Fibrosis; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual, group CF-CBT (Experimental)
  Interventions: Behavioral: Virtual, Group CF-CBT

INTERVENTIONS:
Behavioral: Virtual, Group CF-CBT — Virtual, group CF-CBT is an online, tailored CBT program for adults diagnosed with CF. Participants will attend eight weekly sessions (90 minutes each) delivered online. The sessions include: Introduction to CBT; Relaxation Skills; Depression in CF: What Helps?; Adaptive Thinking Skills, Part 1; Adaptive Thinking Skills, Part 2; Taking Charge of My Health; Anxiety in CF: What Helps?; and Maintaining Positive Changes.

SUMMARY:
The overall goal of this clinical trial is to: a) explore the feasibility, acceptability, and participant experiences with the group version of CF-CBT; b) examine the effectiveness of the virtual delivery of a group version of CF-CBT in reducing depression and anxiety symptoms, perceived stress, coping skills, and health related quality of life among adults with CF.

The primary research questions is:

• How feasible and acceptable (i.e., drop out, adherence, and satisfaction) is virtual, group CF-CBT?

The secondary research questions is:

• How will virtual, group CF-CBT affect depression and anxiety?

The tertiary/other research questions are:

* How will virtual, group CF-CBT affect perceived stress, coping skills, and health related quality of life?
* What is the association between group cohesion and depression, anxiety, perceived stress, coping skills, and health related quality of life?

Participants will:

* Complete short demographic questionnaire regarding their personal and health information.
* Complete questionnaires about symptoms of depression, anxiety, perceived stress, coping skills, and health related quality of life at pre- and post-program. An additional measure of treatment expectancy will be completed at pre-program only. At post-program only, measures of group cohesion and treatment satisfaction will be completed.
* Complete the CF-CBT online mental health program over eight weeks.
* Be invited to complete an interview about their experiences with the program.

Primary outcomes will be compared to benchmark study of individual CF-CBT. Secondary outcomes (i.e., depression, anxiety) will be compared against themselves (i.e., pre- and post-group). Tertiary/other outcomes (i.e., perceived stress, coping skills, health related quality of life) will be compared against themselves (i.e., pre- and post-group). The associations between self-reported outcome measures and group cohesion will be analyzed by computing Pearson correlation coefficients.

DETAILED DESCRIPTION:
BACKGROUND: CF is a genetic, life-limiting, chronic disease that affects approximately 4300 Canadians (~70,000 to 100,000 patients worldwide; Cystic Fibrosis Canada, 2018; Cystic Fibrosis Worldwide, n.d.; Sawicki et al., 2011). People with cystic fibrosis (pwCF) demonstrate high rates of depression and anxiety (Quittner et al., 2014) and the corresponding deleterious impact on functioning is alarming (e.g., decreased lung function and worse adherence to critical life prolonging therapies; Smith et al., 2010; Yohannes et al., 2012). While evidence-based psychological approaches for depression and anxiety, such as cognitive behavioral therapy (CBT), are effective in reducing depression and anxiety symptoms that are co-morbid with other chronic illnesses (e.g., diabetes, COPD, and cancer; Uchendu & Blake, 2016; Williams et al., 2020; Shi et al., 2019; Gandy et al., 2013; López-López et al., 2019), there is a need to design tailored treatments to address the specialized needs of pwCF. To this end, Friedman, Georgiopoulos, and colleagues developed CF-CBT, an innovative, effective, 8-session, individually delivered CF-specific CBT-based intervention program to promote emotional well-being for adults with CF (Friedman et al., 2022a; Friedman et al., 2022b). Virtual delivery of CF-CBT in a group format is one way to address the potentially prohibitive costs of mental health treatment while also addressing infection control guidelines for pwCF, which preclude in-person groups (Saiman et al., 2014)). CF-CBT has been recently modified (i.e., session structure, activities) for group delivery; however, feasibility, acceptability, effectiveness of, and patient experiences with this mode of delivery have yet to be investigated.

PARTICIPANTS: G*Power 3.1 was used to calculate the study sample size based upon on secondary analyses (i.e., t-test). Assuming 80% power, an alpha of 0.05, and an effect size of 0.5 (medium), a sample size of at least 27 participants would be needed. The investigation aims to recruit 28-30 participants to address attrition. Participants with CF will be recruited from CF clinics in British Columbia, Canada. Participants will be consecutively enrolled into groups upon completing pre-program measures. The investigators will seek to have a 2:1 women to men ratio to address gender variations in mental health symptoms and disorders.

HYPOTHESES:

Primary hypothesis:

1. Virtual, group CF-CBT will be feasible and acceptable, as indexed by low rates of drop out and high rates of adherence and satisfaction.

   Secondary hypothesis:
2. There will be significant improvements in self-reported depression and anxiety from pre- to post-program.

   Tertiary/other hypotheses:
3. There will be significant improvements in self-reported perceived stress, coping skills, and health related quality of life from pre- to post-program.
4. Self-reported group cohesion will be negatively associated with depression, anxiety, perceived stress, coping skills, and health related quality of life at post-program.

METHODS/PROCEDURES: Participants with mild-moderate anxiety and/or depression (as measured by the GAD-7 and PHQ-9) (as identified in routine mental health screeing in CF clinic) will be provided information on the study. Those interested in participating will have their email sent to the primary investigator (PI). The PI will email interested participants with a link to Qualtrics, containing the consent form, demographics form, and pre-program questionnaires to be completed before starting the program. Consecutively enrolled participants will be assigned to a virtual CF-CBT group (6-8 participants/group), with the group running for 90 minutes per week over eight weeks. Weekly sessions will be delivered virtually by two trained facilitators (clinical social workers) on the healthcare version of Zoom. Rates of participant enrollment and attrition will be recorded and a treatment fidelity checklist will be completed for 20% of sessions in real-time (by research assistant). Upon completion of the program, participants will be emailed by the PI with another Qualtrics link for the post-program questionnaires.

ANALYSES: Analyses will be completed using IBM SPSS Statistics-Version 26. Demographic and feasibility data (i.e., enrollment and attrition), and measure total scores will be reported (i.e., means and standard deviations for continuous data, frequencies and percentages for categorical data). Primary analyses: The primary outcomes will be compared to benchmark study of individual CF-CBT. Secondary analyses: Secondary outcomes will be analyzed using paired t-tests. Cohen's d metric of effect sizes (ES) of pre-post mean change scores will be used to assess the magnitude of the effects. Tertiary/other analyses: Tertiary/other outcomes will be analyzed using paired t-tests. Cohen's d metric of effect sizes (ES) of pre-post mean change scores will be used to assess the magnitude of the effects. The associations between self-reported outcome measures and group cohesion will be analyzed by computing Pearson correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Must speak and read in English.
* Must have depression and/or anxiety scores in the mild to moderate range (as per the PHQ-9 and GAD-7) prior to study baseline.

Exclusion Criteria:

* Those with suicidal intent (either with or without a plan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of virtual group CF-CBT. | From recruitment to completion of treatment (8 weeks).
  Determined by rates of program completion and program satisfaction.
Feasibility of virtual, group CF-CBT. | From recruitment to completion of treatment (8 weeks).
  Determined by rates of participants recruitment (i.e., how many are interested, enroll) and rates of attendance.
Participant scores on the Client Satisfaction Questionnaire (CSQ) at the end of 8 week treatment. | Post-intervention (8 weeks)
  The CSQ measures satisfaction with a received service on an 8-item scale with items reflecting how satisfied the individual was with the service they completed. Total scores can range from a minimum score of 8 to a maximum score of 32.

SECONDARY OUTCOMES:
Change from baseline in the Patient Health Questionnaire-9 (PHQ-9) at the end of 8 week treatment. | Baseline and post-intervention (8 weeks)
  The PHQ-9 is a measures depression on a 9-item scale with items being rated on a 4-point Likert scale reflecting frequency of depressive symptoms. Total scores can range from a minimum score of 0 to a maximum score of 27.
Change from baseline in the Generalized Anxiety Disorder-7 (GAD-7) at the end of 8 week treatment. | Baseline and post-intervention (8 weeks)
  The GAD-7 measures anxiety on a 7-item scale with items being rated on a 4-point Likert scale reflecting the frequency of anxiety symptoms. Total scores can range from a minimum score of 0 to a maximum score of 21.

OTHER OUTCOMES:
Change from baseline in the Perceived Stress Scale (PSS) at the end of 8 week treatment. | Baseline and post-intervention (8 weeks)
  The PSS measures perceived stress on a 14-item scale with items being rated on a 5-point Likert scale reflecting frequency of perceived stress. Total scores can range from a minimum score of 0 to a maximum score of 56.
Change from baseline in the CF coping self-efficacy scale (CF-CSE) at the end of 8 week treatment. | Baseline and post-intervention (8 weeks)
  The CF-CSE measures CF coping skills on a 21-item scale with items being rated on scale of 10-100 reflecting confidence in ability to cope. Total scores can range from a minimum score of 210 to a maximum score of 2100.
Change from baseline in the Cystic Fibrosis Questionnaire - Revised (CFQ-R) at the end of 8 week treatment. | Baseline and post-intervention (8 weeks)
  The CFQ-R measures health related quality of life for individuals with CF on a 44-item scale with items being rated on 4-point Likert scale reflecting how much CF has impacted one's life. Total scores can range from a minimum score of 44 to a maximum score of 176.
Participant scores on the Group Cohesion Scale - Revised (GCS-R) at the end of 8 week treatment. | Post-intervention (8 weeks)
  The GCS-R measures group cohesion on a 25-item scale with items being rated on 4-point Likert scale reflecting the connections the individual had with other group members. Total scores can range from a minimum score of 25 to a maximum score of 100.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Paul Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia